CLINICAL TRIAL: NCT03652909
Title: Personal Sound Amplification Smartphone Application Feasibility Study
Brief Title: Personal Sound Amplification Smartphone Application Feasibility
Acronym: PSAD
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Wisconsin, Milwaukee (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO00032080; R41DC017939 (NIH)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with difficulty hearing in some daily listening situations: Patients listen to sounds with and without the personal sound amplification smartphone application
  Interventions: Device: Ascending Hearing Technologies device

INTERVENTIONS:
Device: Ascending Hearing Technologies device — Personal Sound Amplification Device

SUMMARY:
Find a personal sound amplification device that can help people hear better.

DETAILED DESCRIPTION:
Personal sound amplification devices (PSADs) have recently become available to the public. PSADs serve a potentially important role in providing audibility of sounds for adults who find themselves having difficulty hearing and understanding speech in some daily living situations, but may not be candidates for traditional, high-amplification hearing aids. Despite hearing loss being a very common problem, few adults who could benefit from some level of amplification actually access the technology. Only approximately 1 in 7 adults (14%) over the age of 50 with a hearing loss using amplification. High cost is the most commonly cited reason for not wanting to try amplification, and indeed, hearing aids range from $1000 to $5000 each (i.e., per ear). PSADs range from $50-$600 each, and may provide a reasonable option for people who are not ready, or are unwilling, to wear a hearing aid. This project aims to examine the feasibility of a PSAD to provide audible and clear sound signal to adult listeners. The significance of this project is its potential to develop an option for individuals to take advantage of amplification and access sound to improve quality of life, who may not otherwise do so without this technology.

ELIGIBILITY:
Inclusion Criteria:

* Adults who report difficulty hearing in some daily listening situations.
* Primarily English-speaking
* Able to follow instructions and perform study procedures.

Exclusion Criteria:

* Children
* Non-English speaking
* Unable to perform research procedures and/or follow necessary instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who report difficulty hearing in some daily listening situations
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Runge, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred February through September 2021. Participants were recruited from the audiology and ear nose and throat clinics.
Pre-assignment Details: Not applicable. Enrollment and subject participation in the experiment occurred sequentially within the same study visit.
Groups:
- PSAD: Patients try the personal sound amplification device.
  Ascending Hearing Technologies device: Personal Sound Amplification Device
Period: Overall Study
Arm/Group | PSAD
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PSAD
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 21
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 62.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
Speech perception percent correct [Mean (Standard Deviation); unit: percent words correct] — Speech perception score is calculated as the percent of words heard correctly
  percent words correct | 57 (34)
Sound quality: Words were clear [Mean (Standard Deviation); unit: score on a scale] — Sound quality was measured using a Likert scale. The Likert rating scale measures the subject's perception of how well she/he heard both with the Personal Sound Amplification Device and without the device. The patient rates the following questions on a scale from Strongly Disagree (value=0), Disagree (value=1), Neutral (value=2), Agree (value=3), and Strongly Agree (value=4) for the statement 'words sounded clear.' Higher values mean better sound quality outcome.
  score on a scale | 1.5 (1.2)
Sound quality: Sentences were easy to understand [Mean (Standard Deviation); unit: score on a scale] — Sound quality was measured using a Likert scale. The Likert rating scale measures the subject's perception of how well she/he heard both with the Personal Sound Amplification Device and without the device. The patient rates the following questions on a scale from Strongly Disagree (value=0), Disagree (value=1), Neutral (value=2), Agree (value=3), and Strongly Agree (value=4) for the statement 'sentences were easy to understand.' Higher values mean better sound quality outcome.
  score on a scale | 1.4 (1.0)
Sound quality: sounds were distorted [Mean (Standard Deviation); unit: score on a scale] — Sound quality was measured using a Likert scale. The Likert rating scale measures the subject's perception of how well she/he heard both with the Personal Sound Amplification Device and without the device. The patient rates the following questions on a scale from Strongly Disagree (value=0), Disagree (value=1), Neutral (value=2), Agree (value=3), and Strongly Agree (value=4) for the statement 'sounds were distorted.' Lower values mean better sound quality outcome.
  score on a scale | 2.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Sentence Perception in Noise Fine-tuned v Unamplified
Description: The fine-tuned Personal Sound Amplification Device sound output will show speech perception benefit over the unamplified condition. Measure is percent of words heard correctly.
Time Frame: The patient will wear the Personal Sound Amplification Device for approximately 30 minutes
Population: All subjects
Measure: Mean (Standard Deviation); unit: percentage of words heard correctly
Groups:
- Personal Amplification: Patients try the personal sound amplification device.
  Ascending Hearing Technologies device: Personal Sound Amplification Device
Arm/Group | Personal Amplification
Number analyzed (Participants) | 32
percentage of words heard correctly | 78 (20)

2. Primary Outcome: Sentence Perception in Noise Initial Fit v Unamplified
Description: The prescription gain (initial fit) Personal Sound Amplification Device sound output will show speech perception benefit over the unamplified condition. Measure is percent of words heard correctly.
Time Frame: The patient will wear the Personal Sound Amplification Device for approximately 30 minutes
Population: All subjects
Measure: Mean (Standard Deviation); unit: percentage of words heard correctly
Groups:
- Personal Amplifier: Patients try the personal sound amplification device.
  Ascending Hearing Technologies device: Personal Sound Amplification Device
Arm/Group | Personal Amplifier
Number analyzed (Participants) | 32
percentage of words heard correctly | 83 (18)

3. Secondary Outcome: Words Clear
Description: The Likert Scale rating scale measures the subject's perception of how well he/she heard both with the Personal Sound Amplification Device and without the device.
  The patient will rate the following questions on a scale from Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), and Strongly Agree (4) for the statement 'the words were clear.' Higher values mean better outcome.
Time Frame: The patient will wear the personal sound amplification device on average for 30 minutes.
Population: All subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personal Amplifier
Number analyzed (Participants) | 32
score on a scale | 2.6 (0.9)

4. Secondary Outcome: Sentences Easy to Understand
Description: The Likert Scale rating scale measures the subject's perception of how well he/she heard both with the Personal Sound Amplification Device and without the device.
  The patient will rate the following questions on a scale from Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), and Strongly Agree (4) for the statement 'sentences were easy to understand.' Higher values mean better outcome.
Time Frame: The patient will wear the Personal Sound Amplification Device for approximately 30 minutes
Population: All subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personal Amplifier
Number analyzed (Participants) | 32
score on a scale | 2.5 (1.1)

5. Secondary Outcome: Sounds Are Distorted
Description: The patient will rate the following questions on a scale from Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), and Strongly Agree (4) for the statement 'the words were clear.' Lower values mean better outcome.
Time Frame: The patient will wear the Personal Sound Amplification Device for approximately 30 minutes
Population: All subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personal Amplifier
Number analyzed (Participants) | 32
score on a scale | 1.6 (1.0)

ADVERSE EVENTS:
Time Frame: 90 minutes
Arm/Group | PSAD
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03652909/Prot_SAP_ICF_000.pdf